CLINICAL TRIAL: NCT05348005
Title: A Cross-Over Study of the Use of Transcutaneous Electrical Nerve Stimulation Unit in the Management of Endometriosis Pain
Brief Title: Use of TENS Unit in the Management of Endometriosis Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kristin Riley, MD, Assistant Professor, Obstetrics and Gynecology; Interim Chief, Minimally Invasive Gynecologic Surgery; Fellowship Program Director, Minimally Invasive Gynecologic Surgery, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00019024
Record Dates: First submitted 2021-12-08; First posted 2022-04-27 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Endometriosis; Pelvic Pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: cross-over clinical study to evaluate the effectiveness of TENS units on the management of endometriosis flare-related pain. Subjects will participate in a 3-month "baseline" period (no TENS unit use for endometriosis flares) and then cross-over to a 3-month "treatment" period (TENS unit use for endometriosis flares).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No TENS unit use (No Intervention): All subjects will start with 3 months of no TENS use and diary tracking
- TENS unit use (Active Comparator): All subjects will then have 3 months of TENS use during episodes of endometriosis pain flare and diary tracking.
  Interventions: Device: Ovira Transcutaneous Electrical Nerve Stimulation Unit

INTERVENTIONS:
Device: Ovira Transcutaneous Electrical Nerve Stimulation Unit — TENS units have a wide application from treatment of chronic back pain, chronic abdominal pain, cancer pain, perioperative pain, and labor pain.19-24 TENS units have been shown to be well-tolerated with minimal side effects and have been successful in reducing pain as well as pain medication use in patients with primary dysmenorrhea, which excludes pathology such as endometriosis. 11-18 Certain TENS units have also been FDA approved for the general indication of pelvic pain.
  Arms: TENS unit use

SUMMARY:
The purpose of this study is see if Transcutaneous Electrical Nerve Stimulator (TENS) units help decrease endometriosis flare pain. TENS units have a 510K and are intended for relief of pain associated with sore or aching muscles of the lower back, arms, or legs due to strain from exercise or normal household and work activities.

Participants will complete surveys, record pain, medication use and bleeding in an online diary during endometriosis flare ups for 3 months without using the TENS unit. After the first 3 month period of time, a TENS unit will be given to participants to wear and again, record pain, medication use and bleeding in the online diary during endometriosis flare ups for and additional 3 months while using the TENS unit.

DETAILED DESCRIPTION:
The investigators propose to conduct a cross-over clinical study to evaluate the effectiveness of TENS units on the management of endometriosis flare-related pain. Subjects will participate in a 3-month "baseline" period (no TENS unit use for endometriosis flares) and then cross-over to a 3-month "treatment" period (TENS unit use for endometriosis flares).

Potential subjects will be pre-screened in the Penn State Minimally Invasive GYN (MIGS) Surgery Clinic for pathologically diagnosed endometriosis and from the Penn State MIGS endometriosis database. Potential subjects will then be called to evaluate the remainder of the inclusion and exclusion criteria. If fulfilled, potential subjects will follow up at the enrollment visit (Visit 1) where consent is reviewed and signed. The baseline QOL and FSFI REDCap surveys will be completed at this visit. Subjects will be set up to receive automated links to complete diary entries and surveys directly in REDCap.

Prior to initiating TENS unit use for endometriosis flare-related pain, subjects will record daily entries into RedCap during episodes of endometriosis flares for 3 months. Each entry will record their VAS pain score as well as medication intake and bleeding profile.

Subjects will then be mailed the TENS unit at the 3 months mark into the study. Subjects will then complete entries with TENS use at their discretion for the following 3 months and record TENS unit use duration, frequency, and side effects in addition to the documentation of pain, medication and bleeding. At the end of the study, subjects will complete a QOL and FSFI survey.

ELIGIBILITY:
Inclusion Criteria:

1. Females ages 18-45 years at time of enrollment
2. A surgical diagnosis with direct visualization and/or histopathologic confirmation of endometriosis
3. Average monthly endometriosis pain flare
4. Naïve TENS user

Exclusion Criteria:

1. TENS device exclusion:

   1. Implantable devices (pacemaker, Interstim, etc.)
   2. Cardiac arrhythmia
   3. Open skin sores over areas of placement
2. Pregnancy
3. Nursing or trying to conceive at this time
4. Post-operative <12 weeks from abdominal or pelvic surgery
5. Planned surgery or hormonal medication changes for duration of study if applicable
6. Non-English speaking or inability to read and understand English
7. Prisoners

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Average Daily VAS Pain Score | Baseline Period (months 1-3) and Treatment Period (months 4-6)
  Average daily pain during endometriosis flares will be measured using a Visual Analog Scale (VAS), a horizontal line measuring pain from 0 (no pain) to 100 (worst pain), and compared between the baseline period (no TENS use) and treatment period (TENS use).

SECONDARY OUTCOMES:
Change in Quality of Life Score from baseline to end of study using the EHP30 questionnaire | Baseline and 6 months
  Change in quality of life from baseline to end of study using the Endometriosis Health Profile (EHP30) questionnaire. Scores range from 0 (best health status) to 100 (worst health status).
Change in Female Sexual Function Index Total Score using the FSFI questionnaire | Baseline and 6 months
  Change in Female Sexual Function Index (FSFI) validated survey scores from baseline to end of study among participants who are currently partnered. FSFI total score ranges from 2.0 (poor) to 36.0 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin W Riley, MD, Principal Investigator — Penn State Health Hershey Medical Center
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burney RO, Giudice LC. Pathogenesis and pathophysiology of endometriosis. Fertil Steril. 2012 Sep;98(3):511-9. doi: 10.1016/j.fertnstert.2012.06.029. Epub 2012 Jul 20. PMID 22819144
- [Result] Bai HY, Bai HY, Yang ZQ. Effect of transcutaneous electrical nerve stimulation therapy for the treatment of primary dysmenorrheal. Medicine (Baltimore). 2017 Sep;96(36):e7959. doi: 10.1097/MD.0000000000007959. PMID 28885348
- [Result] Giudice LC, Kao LC. Endometriosis. Lancet. 2004 Nov 13-19;364(9447):1789-99. doi: 10.1016/S0140-6736(04)17403-5. PMID 15541453
- [Result] Lamvu G, Soliman AM, Manthena SR, Gordon K, Knight J, Taylor HS. Patterns of Prescription Opioid Use in Women With Endometriosis: Evaluating Prolonged Use, Daily Dose, and Concomitant Use With Benzodiazepines. Obstet Gynecol. 2019 Jun;133(6):1120-1130. doi: 10.1097/AOG.0000000000003267. PMID 31135725
- [Result] Coxon L, Horne AW, Vincent K. Pathophysiology of endometriosis-associated pain: A review of pelvic and central nervous system mechanisms. Best Pract Res Clin Obstet Gynaecol. 2018 Aug;51:53-67. doi: 10.1016/j.bpobgyn.2018.01.014. Epub 2018 Feb 15. PMID 29525437
- [Result] Rocha MG, e Silva JC, Ribeiro da Silva A, Candido Dos Reis FJ, Nogueira AA, Poli-Neto OB. TRPV1 expression on peritoneal endometriosis foci is associated with chronic pelvic pain. Reprod Sci. 2011 Jun;18(6):511-5. doi: 10.1177/1933719110391279. Epub 2010 Dec 15. PMID 21160085
- [Result] O'Hara R, Rowe H, Fisher J. Self-management in condition-specific health: a systematic review of the evidence among women diagnosed with endometriosis. BMC Womens Health. 2019 Jun 19;19(1):80. doi: 10.1186/s12905-019-0774-6. PMID 31216998
- [Result] Armour M, Sinclair J, Chalmers KJ, Smith CA. Self-management strategies amongst Australian women with endometriosis: a national online survey. BMC Complement Altern Med. 2019 Jan 15;19(1):17. doi: 10.1186/s12906-019-2431-x. PMID 30646891
- [Result] Goncalves AV, Makuch MY, Setubal MS, Barros NF, Bahamondes L. A Qualitative Study on the Practice of Yoga for Women with Pain-Associated Endometriosis. J Altern Complement Med. 2016 Dec;22(12):977-982. doi: 10.1089/acm.2016.0021. Epub 2016 Aug 23. PMID 27552065
- [Result] Huijs E, Nap A. The effects of nutrients on symptoms in women with endometriosis: a systematic review. Reprod Biomed Online. 2020 Aug;41(2):317-328. doi: 10.1016/j.rbmo.2020.04.014. Epub 2020 May 15. PMID 32600946
- [Result] Leonardi M, Horne AW, Vincent K, Sinclair J, Sherman KA, Ciccia D, Condous G, Johnson NP, Armour M. Self-management strategies to consider to combat endometriosis symptoms during the COVID-19 pandemic. Hum Reprod Open. 2020 Jun 1;2020(2):hoaa028. doi: 10.1093/hropen/hoaa028. eCollection 2020. PMID 32509977
- [Result] Schiotz HA, Jettestad M, Al-Heeti D. Treatment of dysmenorrhoea with a new TENS device (OVA). J Obstet Gynaecol. 2007 Oct;27(7):726-8. doi: 10.1080/01443610701612805. PMID 17999304
- [Result] Vance CG, Dailey DL, Rakel BA, Sluka KA. Using TENS for pain control: the state of the evidence. Pain Manag. 2014 May;4(3):197-209. doi: 10.2217/pmt.14.13. PMID 24953072
- [Result] Lauretti GR, Oliveira R, Parada F, Mattos AL. The New Portable Transcutaneous Electrical Nerve Stimulation Device Was Efficacious in the Control of Primary Dysmenorrhea Cramp Pain. Neuromodulation. 2015 Aug;18(6):522-6; discussion 522-7. doi: 10.1111/ner.12269. Epub 2015 Feb 5. PMID 25655828
- [Result] Machado AFP, Perracini MR, Rampazo EP, Driusso P, Liebano RE. Effects of thermotherapy and transcutaneous electrical nerve stimulation on patients with primary dysmenorrhea: A randomized, placebo-controlled, double-blind clinical trial. Complement Ther Med. 2019 Dec;47:102188. doi: 10.1016/j.ctim.2019.08.022. Epub 2019 Aug 28. PMID 31779988
- [Result] Igwea SE, Tabansi-Ochuogu CS, Abaraogu UO. TENS and heat therapy for pain relief and quality of life improvement in individuals with primary dysmenorrhea: A systematic review. Complement Ther Clin Pract. 2016 Aug;24:86-91. doi: 10.1016/j.ctcp.2016.05.001. Epub 2016 May 7. PMID 27502806
- [Result] Kannan P, Claydon LS. Some physiotherapy treatments may relieve menstrual pain in women with primary dysmenorrhea: a systematic review. J Physiother. 2014 Mar;60(1):13-21. doi: 10.1016/j.jphys.2013.12.003. Epub 2014 Apr 24. PMID 24856936
- [Result] Greco CD. Management of adolescent chronic pelvic pain from endometriosis: a pain center perspective. J Pediatr Adolesc Gynecol. 2003 Jun;16(3 Suppl):S17-9. doi: 10.1016/s1083-3188(03)00064-0. PMID 12742182
- [Result] Sluka KA, Bjordal JM, Marchand S, Rakel BA. What makes transcutaneous electrical nerve stimulation work? Making sense of the mixed results in the clinical literature. Phys Ther. 2013 Oct;93(10):1397-402. doi: 10.2522/ptj.20120281. Epub 2013 May 2. PMID 23641031
- [Result] Harvey MP, Watier A, Dufort Rouleau E, Leonard G. Non-invasive stimulation techniques to relieve abdominal/pelvic pain: Is more always better? World J Gastroenterol. 2017 May 28;23(20):3758-3760. doi: 10.3748/wjg.v23.i20.3758. PMID 28611529
- [Result] Dowswell T, Bedwell C, Lavender T, Neilson JP. Transcutaneous electrical nerve stimulation (TENS) for pain relief in labour. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007214. doi: 10.1002/14651858.CD007214.pub2. PMID 19370680
- [Result] Hurlow A, Bennett MI, Robb KA, Johnson MI, Simpson KH, Oxberry SG. Transcutaneous electric nerve stimulation (TENS) for cancer pain in adults. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD006276. doi: 10.1002/14651858.CD006276.pub3. PMID 22419313
- [Result] Johnson MI. Transcutaneous electrical nerve stimulation (TENS) as an adjunct for pain management in perioperative settings: a critical review. Expert Rev Neurother. 2017 Oct;17(10):1013-1027. doi: 10.1080/14737175.2017.1364158. Epub 2017 Aug 24. PMID 28817978
- [Result] Proctor ML, Smith CA, Farquhar CM, Stones RW. Transcutaneous electrical nerve stimulation and acupuncture for primary dysmenorrhoea. Cochrane Database Syst Rev. 2002;2002(1):CD002123. doi: 10.1002/14651858.CD002123. PMID 11869624